CLINICAL TRIAL: NCT01420900
Title: Ceramic-on-Ceramic Total Hip Arthroplasty and Squeaking: A Prospective, Blinded, Randomized Clinical Trial of Influence of Component Design
Brief Title: Ceramic-on-Ceramic Total Hip Arthroplasty and Squeaking: Influence of Component Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Principal Investigator, Claus Varnum, MD, Vejle Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: man2if
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Hip Arthrosis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABG II / Trident (Active Comparator)
  Interventions: Device: THA with ABG II / Trident
- CLS / Trilogy (Active Comparator)
  Interventions: Device: THA with CLS / Trilogy

INTERVENTIONS:
Device: THA with ABG II / Trident — Surgery with total hip arthroplasty in the form of ABG II / Trident
  Arms: ABG II / Trident
Device: THA with CLS / Trilogy — Surgery with total hip arthroplasty in the form of CLS / Trilogy
  Arms: CLS / Trilogy

SUMMARY:
The investigators want to examine if specific acetabular liner designs can be a contributing factor to audible squeaking associated with CoC bearings. The aim of the present study is to compare two different designed and well documented acetabular component systems with reference to squeaking and other noises from the hip.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for uncemented THA under the age of 65 years.

Exclusion Criteria:

* Patients with the following diagnoses of the hip: Recent femoral fracture, sequelae from older femoral fracture, acetabular fracture, and traumatic dislocation of the hip.
* Patients without ability to give informed consent and/or willingness to participate in the follow-up protocol.
* Severely impaired level of function due to other physical deficiencies than the hip.
* Mental disability that could impair a patient's decision-making capability of giving informed consent and not enabling valid data collection.
* Earlier primary THA or revision THA in the contralateral hip.
* Pathology requiring another prosthesis concept than the below mentioned.
* Body mass index greater than 35.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2011-09; Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
All noises from THA | One year

SECONDARY OUTCOMES:
Life quality | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedic Surgery, Vejle Hospital, Vejle, Denmark